CLINICAL TRIAL: NCT04123769
Title: Pharmacokinetics of Hydronidone Capsules in Patients With Chronic Hepatitis B Complicated With Liver Fibrosis and Mild Hepatic Insufficiency
Brief Title: Study on PK of Hydronidone in Patients and Special Population
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GNI-F351-201901
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Hepatitis b & Liver Dysfunction
MeSH Terms: conditions — Hepatitis B; Liver Diseases | interventions — hydronidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug group (Experimental)
  Interventions: Drug: Hydronidone

INTERVENTIONS:
Drug: Hydronidone — First take Hydronidone capsule, single-dose and then Multiple-dose

SUMMARY:
1. Evaluate the pharmacokinetic (PK) characteristics of Hydronidone capsule in target patients (patients with chronic viral hepatitis b with liver fibrosis) and special population (patients with mild liver dysfunction).
2. To evaluate the effect of oral Hydronidone capsule on QT/QTc in patients with chronic viral hepatitis b accompanied by hepatic fibrosis and mild hepatic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years (including 18 and 65 years);
2. BMI 18-26 (including 18 and 26) [BMI= weight (kg)/height 2 (m2)];
3. History of chronic hepatitis b, HBsAg positive ≥6 months;
4. ALT < 5 times ULN (standard upper limit);
5. TBiL < 2 times ULN (standard upper limit);
6. ALP < 1.5 times ULN (standard upper limit);
7. Liver elastic hardness test confirmed significant liver fibrosis (LSM≥ 7.3kpa);
8. Scores assessed by child-pugh system are 5 or 6;
9. Patients currently receiving antiviral treatment with entecavir;
10. The subject (or his/her partner) has no pregnancy plan during and within 6 months after the trial and voluntarily takes effective physical contraception and has no sperm or egg donation plan;
11. Before the trial, I have had a detailed understanding of the nature, significance, possible benefits, possible inconveniences and potential risks of the trial, and I have volunteered to participate in the clinical trial. I am able to communicate well with the investigator, comply with the requirements of the whole study, and have signed a written informed consent.

Exclusion Criteria:

1. Those who do not meet any of the inclusion criteria;
2. (consultation) participants in clinical trials of other drugs in recent 3 months;
3. (consultation) any drugs that inhibit or induce drug metabolism in the liver (common liver enzyme inducers: barbiturates (phenobarbital is the most common), carbamazepine, aminoximate, griseofulvin, aminopropyl ester, phenytoin, gromitol, rifampin, dexamethasone; Common liver enzyme inhibitors: chlorpromazine, cimetidine, ciprofloxacin, metronidazole, chloramphenicol, isoniazid, sulfonamide);
4. (consultation) select those who drank excessive amounts of tea, coffee or caffeinated beverages (more than 8 cups a day, 1 cup =250mL) every day during the first three months; Or from the screening to -1 days after admission, intake of any food or drink containing caffeine and xanthine (such as coffee, strong tea, chocolate, etc.) and other special diet that affects the absorption, distribution, metabolism and excretion of drugs;
5. (consultation) patients who had taken food or drinks containing enzymes that can induce or inhibit liver metabolism (e.g., grapefruit, mango, pitaya, grape juice, orange juice and other compounds rich in flavonoids or citrus glycosides) before admission were screened.
6. (consultation) screening: drinking more than 14 standard units of alcohol per week in the first 3 months (1 standard unit contains 14g of alcohol, such as 360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine); Or cannot abstain from alcohol during the test period; Or taking any alcohol products within 24 hours before the first dose of the study;
7. (consultation) select those who smoke more than 5 cigarettes per day within the first 3 months, or cannot stop using any tobacco products during the trial; Screening for smoking or using any tobacco products up to admission;
8. (consultation) previous history of drug abuse and drug abuse;
9. (consultation) patients with upper gastrointestinal massive bleeding or active peptic ulcer within the first 3 months were enrolled;
10. (consultation) patients with serious diseases of cardiovascular, pulmonary, renal, endocrine, nervous and blood systems and mental disorders;
11. (consultation) allergy: if allergic to two or more drugs or food; Lactose intolerant;
12. AFP > 100 μg /L;
13. B ultrasound showed obvious space-occupying lesions in the liver, suggesting tumor;
14. Patients with decompensated liver cirrhosis;
15. Patients with malignant tumors;
16. Received non-entecavir nucleoside analogues or interferon antiviral therapy within 3 months before inclusion;
17. Pregnant and/or lactating women;
18. Subjects who are legally disabled according to the law of the People's Republic of China on the protection of disabled persons (April 2008);
19. Alcohol breath test results greater than 0.0mg/100mL;
20. Positive urine drug screening;
21. Patients with suspected poor compliance;
22. The investigator considers that there are any circumstances that may affect the subject's informed consent or adherence to the study protocol, or participation in the study may affect the results of the study or their own safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 24 weeks
Tmax | up to 24 weeks
AUC | up to 24 weeks
QT/QTc | up to 24 weeks

SECONDARY OUTCOMES:
CL/F | up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Medical ethics committee of wuhan infectious disease hospital, Wuhan, Hubei, China